CLINICAL TRIAL: NCT02236624
Title: Can Aerobic Exercise Reduce Flu-like Symptoms Following Interferon Beta 1a Injections in Patients With Multiple Sclerosis?
Brief Title: Aerobic Exercise and Flu-like Symptoms Following Interferon Beta 1a Injections in Patients With Multiple Sclerosis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); MS-Clinic of Southern Jutland (Unknown); MS-Clinic Viborg (Unknown); MS-Clinic Odense (Unknown); Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Avonex
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

ARMS (1):
- Aerobic Exercise (Experimental)
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise

SUMMARY:
The purpose of the present study is to test the hypothesis that aerobic training can reduce flu-like symptoms following interferon beta 1a injections in patients with Multiple Sclerosis.

A secondary purpose is to evaluate whether or not changes in circulating cytokines provide a mechanism that can explain a potential positive effect.

DETAILED DESCRIPTION:
Flu-like symptoms (FLS) such as fever, muscle aches, chills, and fatigue are common side effects of interferon beta (IFN-ß) treatment and may affect the willingness of patients with multiple sclerosis (MS) to initiate therapy. The initiation phase of MS treatment is a critical period that can affect patients' views on the long-term acceptability and the adherence to the therapy, underscoring the need for strategies to reduce treatment-related adverse events such as FLS following IFN-ß injections.

Once-weekly intramuscular IFNß-1a, which has been available since 1996, is indicated for the treatment of patients with relapsing forms of MS to slow the accumulation of physical disability progression and the frequency of clinical exacerbations. Although intramuscular IFNß-1a is generally well tolerated, FLS have been reported in up to 76% of patients receiving this treatment. Consequently, interventions that can reduce FLS after IFNß-1a injection are warranted. One approach to reduce FLS has been dose titration. Titration is the practice of initiating therapy with a lower starting dose and gradually increasing the dose at defined intervals until the full dose is reached. Moreover, a combination of dose titration and pre-treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen in healthy subjects, has been sown to reduce FLS severity by 37-76%. However, not all patients benefit from dose titration and also the effects in MS still have to be determined. Consequently, other types of FLS management after IFNß-1a injection have to be determined.

Interestingly, case reports from both Finland and Denmark suggest that aerobic exercise is able to markedly reduce FLS symptoms in MS patients, but so far no studies have evaluated this. However, from healthy subjects it is known that aerobic exercise is capable of positively influencing the immune system and evidence suggests that the prophylactic effect of exercise may, to some extent, be the induction of an anti-inflammatory environment with each bout of exercise (e.g. via increases in circulating anti-inflammatory cytokines including interleukin (IL)-1 receptor antagonist and IL-10).

The existing evidence is particularly suggestive of an acute effect of aerobic exercise on the circulating cytokine levels, which could be an important mechanism in explaining a potential positive effect of aerobic exercise on FLS.

Consequently, the purpose of the present study is to test the hypothesis that aerobic training can reduce FLS following interferon beta 1a injections in patients with Multiple Sclerosis.

A secondary purpose is to evaluate whether or not changes in circulating cytokines provide a mechanism that can explain a potential positive effect.

ELIGIBILITY:
Inclusion Criteria:

* Definite relapsing-remitting MS according to the McDonald criteria
* Treated with IFNß-1a (Avonex®) for at least 6 months
* Frequent experiencing FLS (muscle aches, chills, fatigue, fewer9) in the hours following IFNß-1a injection (self-reporting that this happens 75% or more of the times after injection).
* Female subjects of childbearing potential are required to practice effective contraception during the study and to continue contraception for 30 days after their last dose of study treatment.
* Expected to be able to complete the aerobic exercise intervention
* Willingly to transport themselves to the exercise/testing facility
* Give informed consent
* Age above 18 years

Exclusion Criteria:

* Have FLS (i.e. muscle aches, chills, fatigue or fewer) or serious infection within a 24h period prior to the screening. Patients having chronic FLS or infection will, therefore, be excluded. This will be tested by patient interview and, if required, further examination
* Have a known history or positive test result for hepatitis B, hepatitis C, or HIV
* Use beta-blockers.
* Have clinically significant abnormality in laboratory or electrocardiogram measures, chronic fatigue syndrome or fibromyalgia, pre-malignant disease, or malignant disease
* Have had allergy shot or desensitization therapy within 1 month of day 1 (randomization) vaccination within 2 weeks of day 1.
* Stop taking IFNß-1a.
* Are pregnant.
* Suffer from dementia, alcohol abuse or have a pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Flu-like symptoms assessment | Change from baseline to 24 hours.
  Comparison of the mean relative change in flu-like symptoms severity from pre-injection to 5 hours post-injection. At 12h and 24h post intervention the participants will further register flu-like symptoms.

SECONDARY OUTCOMES:
Bloodbourne biomarkers | Baseline to 24h
  Bloodbourne biomarkers: Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Martin Langeskov-Christensen, MSc, Principal Investigator — Sport Science, Department of Public Health, Aarhus University; Ulrik Dalgas, PhD, Study Chair — Sport Science, Department of Public Health, Aarhus University; Egon Stenager, Dr.med., Study Chair — MS-Clinic of Southern Jutland (Sønderborg, Vejle, Esbjerg), Department of Neurology, Sønderborg, Denmark and Institute of Regional Health Services, University of Southern Denmark.; Thor Petersen, Dr.med., Study Chair — MS-Clinic Aarhus, Department of Neurology, Aarhus University Hospital, Denmark
Locations (1):
- Sport Science, Department of Public Health, Aarhus University, Aarhus, Aarhus C, Denmark